CLINICAL TRIAL: NCT03305770
Title: DD T2 Daily Disposable Registration Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C005
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Myopia; Refractive Errors
Keywords: soft contact lenses; vision; eyesight
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DD T2 (Experimental): Verofilcon A contact lenses worn in both eyes for 3 months in a daily wear, daily disposable modality. A new pair of study lenses will be inserted each day and discarded at the end of the day.
  Interventions: Device: verofilcon A contact lenses
- DT 1 (Active Comparator): Delefilcon A contact lenses worn in both eyes for 3 months in a daily wear, daily disposable modality. A new pair of study lenses will be inserted each day and discarded at the end of the day.
  Interventions: Device: delefilcon A contact lenses

INTERVENTIONS:
Device: verofilcon A contact lenses — Daily disposable soft contact lenses
  Other Names: DD T2
  Arms: DD T2
Device: delefilcon A contact lenses — Daily disposable soft contact lenses
  Other Names: DAILIES TOTAL1®; DT1
  Arms: DT 1

SUMMARY:
The purpose of this study is to evaluate the performance of the investigational verofilcon A contact lens compared to the commercially available delefilcon A contact lens, by assessing visual acuity as the primary variable.

DETAILED DESCRIPTION:
Enrolled participants will be randomized (2:1) to receive either verofilcon A (test) contact lenses or delefilcon A (control) contact lenses for wear in both eyes and attend 7 office visits: Baseline, Dispense, 1-week follow-up, 2-week follow-up, 1-month follow-up, 2-month follow-up and 3-month follow-up/Exit.

ELIGIBILITY:
Inclusion Criteria:

* Successful wear of spherical soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Best corrected VA 20/25 or better in each eye.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria

* Any current or prior wear experience with DT1 lenses.
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, a Novartis Division, Study Director — Alcon, a Novartis Division
Locations (6):
- United States (6):
  - Alcon Investigative Site, San Diego, California
  - Alcon Investigative Site, Longwood, Florida
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Brentwood, Tennessee
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 investigational sites located in the US.
Pre-assignment Details: This reporting group includes all randomized subjects (107).
Units Other Than Participants: Eyes
Groups:
- DD T2: Verofilcon A contact lenses worn in both eyes for 3 months in a daily wear, daily disposable modality. A new pair of study lenses were inserted each day and discarded at the end of the day.
- DT 1: Delefilcon A contact lenses worn in both eyes for 3 months in a daily wear, daily disposable modality. A new pair of study lenses were inserted each day and discarded at the end of the day.
Period: Overall Study
Arm/Group | DD T2 | DT 1
Started (All randomized subjects) | 70; 140 Eyes | 37; 74 Eyes
Enrolled Dispensed Analysis Set (Enrolled subjects/eyes exposed to study lenses) | 70; 140 Eyes | 36; 72 Eyes
Completed Analysis Set (Subjects/eyes in the Enrolled Dispensed set that completed the study) | 69; 138 Eyes | 36; 72 Eyes
Completed | 69; 138 Eyes | 36; 72 Eyes
Not Completed | 1; 2 Eyes | 1; 2 Eyes
Not completed — Physician Decision - prior to dispense | 0 | 1
Not completed — Subject moved | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis set includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | DD T2 | DT 1 | Total
Number analyzed (Participants) | 70 | 37 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (6.3) | 31.3 (7.6) | 33.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 30 | 81
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 65 | 33 | 98
  Black or African American | 3 | 3 | 6
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1
  Multi-racial | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Visual Acuity (VA) With Contact Lenses at Each Visit (Snellen)
Description: VA was assessed for each eye individually using a Snellen chart at a distance of 4 meters. A 20/20 Snellen acuity is considered normal distance eyesight. No formal hypotheses were formulated; hence no inferential testing was performed.
Time Frame: Dispense, Week 1, Week 2, Month 1, Month 2, Month 3
Population: Completed Analysis Set
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | DD T2 | DT 1
Number analyzed (Participants) | 69 | 36
Number analyzed (eyes) | 138 | 72
eyes
  Dispense @ 20/15 | 74 | 32
  Dispense @ 20/20 | 62 | 40
  Dispense @ 20/25 | 2 | 0
  Dispense @ 20/30 | 0 | 0
  Week 1 @ 20/15 | 75 | 36
  Week 1 @ 20/20 | 58 | 36
  Week 1 @ 20/25 | 4 | 0
  Week 1 @ 20/30 | 1 | 0
  Week 2 @ 20/15 | 69 | 35
  Week 2 @ 20/20 | 65 | 37
  Week 2 @ 20/25 | 4 | 0
  Week 2 @ 20/30 | 0 | 0
  Month 1 @ 20/15 | 62 | 31
  Month 1 @ 20/20 | 72 | 40
  Month 1 @ 20/25 | 4 | 1
  Month 1 @ 20/30 | 0 | 0
  Month 2 @ 20/15 | 63 | 33
  Month 2 @ 20/20 | 68 | 36
  Month 2 @ 20/25 | 7 | 3
  Month 2 @ 20/30 | 0 | 0
  Month 3 @ 20/15 | 63 | 35
  Month 3 @ 20/20 | 69 | 37
  Month 3 @ 20/25 | 6 | 0
  Month 3 @ 20/30 | 0 | 0

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 15 weeks
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Completed Analysis Set. "At Risk" population for ocular AEs is included with unit of "eyes."
Groups:
- DD T2 Ocular: Eyes exposed to verofilcon A contact lenses
- DD T2 Non-ocular: Subjects exposed to verofilcon A contact lenses
- DT 1 Ocular: Eyes exposed to delefilcon A contact lenses
- DT 1 Non-ocular: Subjects exposed to delefilcon A contact lenses
Arm/Group | DD T2 Ocular | DD T2 Non-ocular | DT 1 Ocular | DT 1 Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/69 | 0/72 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/69 | 0/72 | 0/36
Other Adverse Events (participants affected / at risk) | 0/138 | 0/69 | 0/72 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03305770/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03305770/SAP_001.pdf